CLINICAL TRIAL: NCT03159728
Title: Efect of Program Caregivers of With Chronic Diseases
Brief Title: Effectiveness Program Caregivers Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Santander (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 039-2015
Record Dates: First submitted 2017-05-17; First posted 2017-05-19 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-10

CONDITIONS: Chronic Disease
Keywords: Ability Care; Caregiver overload; Family caregiver
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educative intervention (Experimental): Who wish to participate in the program "Caring for Caregivers" will be the intervention group. The intervention or program "Caring for Caregivers" to develop was proposed by the Group of Chronic Care Patient and Family School of Nursing at the National University of Colombia. This program includes four sessions or meetings with the caretaker, induction and three modules, the first is geared to strengthen the knowledge; the second, to strengthen the value and the third, to strengthen patience.
  Interventions: Behavioral: Educative intervention:
- Control group (No Intervention): The control group will receive training about knowledge of chronic disease and care.
  In addition, once it confirmed the effectiveness of the intervention participants in the control group will be contacted to contemplate the possibility of receiving the benefits of the intervention.

INTERVENTIONS:
Behavioral: Educative intervention: — * In the induction of the new group members are present, including caregivers who start the program and those who coordinated.
  * In Module I: to strengthen the knowledge of the situation and the people involved in care.
  * In Module II: to strengthen the value in the caregiver through decision making, skill and social support to back it up.
  * In Module III: or end, after analyzing that uneasy caregiver, patience is reviewed through the meaning of family care and self.
  Arms: Educative intervention

SUMMARY:
In Colombia as in the world, chronic diseases occupy the first places of death being cardiovascular, chronic respiratory diseases and diabetes mellitus are the most prevalent. The caregiver burden is reflected as an experience of constant attention, this routine is shown in the changes they undergo in their life, and the emotions cope at different stages of the process that arises chronic non-communicable disease from their family in demands care. Methodology: a randomized controlled trial (RCT) will be conducted to determine the effect of skill care program "Caring for the caregivers" to reduce the burden of care in carers of people with chronic non-communicable University Hospital in Los Comuneros in Bucaramanga. Results and expected impact: bring to the lines of research: Community Care: improve the ability of the care of family caregivers at home and increase the quality of life that people are able to chronicity. Clinical Care: Strengthens care ability of caregivers who are in health institutions. Management and Care Management: Promoting implementation, monitoring and evaluation of the educational proposal in order to create a network of support for family caregivers in Santander in extending the results to other institutions. The project results should allow participation in Extension and Social Projection, whose results will allow the implementation of an effective educational model for the care of patients with chronic non-communicable disease in Colombia. In addition, the consolidation of the alliance between Everest group at the University of Santander with the Latin American Network of chronic patient care and clinical Communards of Bucaramanga projects. Finally it is expected to consolidate training in the area of research students in undergraduate and graduate programs at the University of Santander.

DETAILED DESCRIPTION:
Chronic noncommunicable diseases (NCDs) are the cause of increased consumption of socio-health resources, this in time and costs of medication these patients, added to this is the aging population that has drawn the attention of economists, politicians, health workers and researchers. At present, the change in the population pyramid is one of the factors that caused the increase in chronic diseases, which are the leading cause of morbidity and mortality worldwide. (Campos, M. Moya, D. Mendoza, D. Child, E., 2014).

The presence of chronic non-communicable diseases makes it of interest of the whole society including the government, private sector and academia, twenty-one making it more advantageous and cost-effective strategies are needed as new media and thus strengthen the capacity of health services to respond to NCDs. (World Health Organization, 2012).

For other part of the (NCCD) usually are long and slow evolution, affecting all age groups and all regions regardless of condition social, besides also they characterized by total or partial loss of autonomy seeing the person who has it must depend wholly or partly from a caregiver who provides security and support during his illness and in the process of recovery, This requires that promote the development of knowledge and skills in people with chronic non-communicable diseases and their caregivers and form social and support networks to facilitate better adaptation process against disease, through sources that allow you to collect systematize and disseminate information in order to improve the level of knowledge and induce changes to behaviors and lifestyles that promote physical and mental health care cuidadorsujeto dyad. (Herrera, A. Florez, I. Romero, E. Montalvo, A. Physical, psychological, social and spiritual implications of chronic non-communicable disease (NCD), affect not only the sufferer, but also their family caregiver (5), which substantiates the need to go beyond the organic approach the same; thus the social support family caregivers of people with NCDs takes importance. (Barrera, L. Campos, M. Carreño, S. Carrillo M, Chaparro,L. Jaimes, M. Ortiz, S. Piratoba, B. Rosales, R. Sánchez, B., 2013) According Colliere quoted by Campos, CARE is an act of life that means an infinite variety of activities to sustain life and enable continuity and reproduction. Garcia says that caring is a habitual simple activity in humans, continually practiced as an integral part of the daily activities of people, to answer the essential aspiration to meet the needs. (Campos, M. Moya, D. Mendoza, D. Child, E., 2014) Escudero says Sitter is "the person or family, which provides most of the care and daily support who suffers from a disease or require assistance for the development of activities of daily living, without receiving financial remuneration" (Campos, M. Moya, D. Mendoza, D. Child, E., 2014) In Colombia in the study by Barreto and collaborators reported that most care for his family since the beginning of the NCCD, with exceeding seven months and more than seven hours per day times, which can mean an oppressive and incompatible work with a good quality of life. However, just over half report not only carers and have braces, spiritual and social family.

Additionally it was found that 8.6% of caregivers reported dysfunction and, particularly, 3.6% reflecting deterioration in mental status, thus the risk of the occurrence of adverse events for themselves and their families with NCDs is very high. (Barreto, R. Campos, M. González, G. Coral, R. Chaparro, L. Duran, M, et al, 2015) This study also found that knowledge and access to information and communication technologies (ICT), mostly middle and upper part, constitute an invaluable opportunity for social support for this group; only 42.8% of caregivers reported healthy.

The results corroborate the charge that the role of caregiver is associated with extensive wear and confirm findings from different studies analyzing the burden of care. (Barreto, R. Campos, M. González, G. Coral, R. Chaparro, L. Duran, M, et al, 2015).

This study adopts the concept of skill care proposed by Nkongho as a multidimensional concept with three dimensions including knowledge, courage and patience. From these principles Nkongho ability develops the concept of care as "the ability to help others grow in a relationship that involves process development." (Eterovic, C. Mendoza, S. Saenz, K. 2015) This project is a research derived "Program Decreased Burden of Chronic Disease Transmissible No (NCDs) in Colombia". In which a pilot test where the results showed the felt need for an educational program on the ability of care in family caregivers of patients with chronic disease was made.

This justifies the realization of this project will allow participation in Extension and Social Outreach, an effective educational model for caregivers of people with non-communicable chronic disease in Colombia. In addition, the consolidation of the alliance between Everest group at the University of Santander with the Latin American Network of chronic patient care and teaching hospital in Bucaramanga The Communards projects. Finally it is expected to consolidate training in the area of research students in undergraduate and graduate programs in specialization in Quality Management and Audit in Health at the University of Santander.

ELIGIBILITY:
Inclusion Criteria:

* Family caregivers of people with chronic non-communicable disease attending the University Hospital Los Comuneros in Bucaramanga.
* Family caregivers for a minimum period of three months
* Be of age

Exclusion Criteria:

* Carers with communication difficulties
* Caregivers difficulty understanding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-06-15 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-03-30 (Estimated)

PRIMARY OUTCOMES:
Care ability | within the first 90 days
  For the measurement of the ability to care Inventory Skill Care (Caring Ability Inventory, CAI) version in Spanish from the original version of Nkongho.

SECONDARY OUTCOMES:
Burden of care | within the first 90 days
  To assess the perception of the burden of care which manages a multidimensional measure the level of care Survey Zarit Burden, an instrument was used caregiver burden perceives its responsibility to care for the person.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia C Torres, RN, MSc, Study Director — Universidad de Santander
Locations (1):
- Santander, Colombia, Bucaramanga, Santander Department, Colombia

IPD SHARING:
Plan to Share IPD: No